CLINICAL TRIAL: NCT02028169
Title: To Observe the Impacts of Anti-TNF's Effectiveness on Improvement in Work Place and Household Productivity for Patients With Psoriatic Arthritis
Brief Title: To Observe the Impacts of Anti-Tumor Necrosis Factor (TNF) Effectiveness on Improvement in Work Place and Household Productivity for Patients With Psoriatic Arthritis (PsA)
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P13-518
Record Dates: First submitted 2014-01-03; First posted 2014-01-07 (Estimated); Results first posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-03

CONDITIONS: Psoriatic Arthritis; Work Productivity
Keywords: Work Productivity; Anti-TNFs; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants Receiving Anti-TNF for PsA: Participants who are actively working (full-time or part-time) with rheumatologist-confirmed PsA for which the physician has initiated treatment with an anti-TNF.

SUMMARY:
This post marketing observational study is designed to provide the initial data on work impairment of PsA patients in Turkey, as well as changes in work impairment, life quality and clinical response during treatment with anti-TNF agents.

ELIGIBILITY:
Inclusion Criteria:

* Actively working, either full-time or part-time
* Previous confirmed diagnosis of PsA by a rheumatologist
* Patients for whom the physician has initiated PsA treatment with an Anti-TNF in accordance with Turkish Ministry of Health regulations and reimbursement criteria
* Able to provide authorization to use and disclose their health related information

Exclusion Criteria:

* Patients with a history of an allergic reaction or significant sensitivity to anti-TNF agents
* Patients with possible follow-up problems during the planned study period or patients who may not be compliant to treatment as evaluated by the investigator/treating physician
* Patients participating in any clinical trial of an experimental drug 30 days prior to the baseline visit

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from both genders will be included to this non-interventional epidemiological study from selected university or state hospitals or Ministry of Health of Turkey training and research hospitals in Turkey.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut Gücük, MD, Study Director — AbbVie

REFERENCES:
- [Derived] Karadag O, Dalkilic E, Ayan G, Kucuksahin O, Kasifoglu T, Yilmaz N, Koca SS, Yazisiz V, Erten PT, Sayarlioglu M, Terzioglu ME, Erten S, Kalyoncu U. Real-world data on change in work productivity, activity impairment, and quality of life in patients with psoriatic arthritis under anti-TNF therapy: a postmarketing, noninterventional, observational study. Clin Rheumatol. 2022 Jan;41(1):85-94. doi: 10.1007/s10067-021-05893-3. Epub 2021 Sep 3. PMID 34477993
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Receiving Anti-TNF for PsA: Participants who are actively working (full-time or part-time) with rheumatologist-confirmed psoriatic arthritis (PsA) for which the physician has initiated treatment with an anti-tumor necrosis factor (TNF).
Period: Overall Study
Arm/Group | Participants Receiving Anti-TNF for PsA
Started | 120
Completed | 92
Not Completed | 28
Not completed — Lost to Follow-up | 21
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1
Not completed — Cessation of Drug | 1
Not completed — Concomitant Medication Usage | 1

BASELINE CHARACTERISTICS:
Arm/Group | Participants Receiving Anti-TNF for PsA
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.65 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 47

OUTCOME MEASURES:

1. Primary Outcome: Work Productivity and Activity Impairment (WPAI) Questionnaire: Mean Percentage of Work Time Missed (Absenteeism) Up to Month 9
Description: Absenteeism, presented as the mean percentage of work time missed due to PsA (as reported on the WPAI), and calculated as: 100*number of hours of work missed due to PsA / (number of hours of work missed due to PsA + number of hours worked). WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity.
Time Frame: Baseline, Month 3, Month 6, Month 9
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Participants Receiving Anti-TNF for PsA
Number analyzed (Participants) | 58
percentage of work time missed
  Baseline | 20.5 (22.2)
  Month 3: number analyzed (Participants) | 48
  Month 3 | 10.0 (20.0)
  Month 6: number analyzed (Participants) | 43
  Month 6 | 7.9 (16.2)
  Month 9: number analyzed (Participants) | 38
  Month 9 | 4.9 (10.5)
Statistical Analysis 1: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 9; Test type: Superiority; p < 0.001, Friedman test

2. Primary Outcome: WPAI Questionnaire: Mean Percentage of Impairment While Working Due to PsA (Presenteeism) Up to Month 9
Description: Presenteeism (the extent to which PsA decreased productivity) is presented as the mean percentage of impairment while working due to PsA, and calculated as: 100*scale value of question 5 on the WPAI (between 0 and 10) / 10. WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity.
Time Frame: Baseline, Month 3, Month 6, Month 9
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: percentage of impairment while working
Arm/Group | Participants Receiving Anti-TNF for PsA
Number analyzed (Participants) | 59
percentage of impairment while working
  Baseline | 53.7 (22.9)
  Month 3: number analyzed (Participants) | 51
  Month 3 | 26.5 (24.1)
  Month 6: number analyzed (Participants) | 46
  Month 6 | 27.1 (24.2)
  Month 9: number analyzed (Participants) | 42
  Month 9 | 19.5 (19.9)
Statistical Analysis 1: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 9; Test type: Superiority; p < 0.001, Friedman test

3. Primary Outcome: WPAI Questionnaire: Mean Percentage of Overall Work Productivity Impairment (OWPI) Due to PsA Up to Month 9
Description: The mean percentage of OWPI due to PsA (based on the WPAI questionnaire) is presented, calculated as: Absenteeism (%) +[1- Absenteeism(%)*Presenteeism(%)]. WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity.
Time Frame: Baseline, Month 3, Month 6, Month 9
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: percentage of OWPI
Arm/Group | Participants Receiving Anti-TNF for PsA
Number analyzed (Participants) | 58
percentage of OWPI
  Baseline | 42.8 (21.4)
  Month 3: number analyzed (Participants) | 48
  Month 3 | 21.6 (18.4)
  Month 6: number analyzed (Participants) | 43
  Month 6 | 21.0 (17.2)
  Month 9: number analyzed (Participants) | 38
  Month 9 | 15.3 (14.2)
Statistical Analysis 1: Comparison: Participants Receiving Anti-TNF for PsA; Baseline Vs. Month 9; Test type: Superiority; p < 0.001, Friedman test

4. Primary Outcome: WPAI Questionnaire: Mean Percentage of Activity Impairment Due to PsA Up to Month 9
Description: Activity impairment due to PsA (the extent to which PsA affected the ability to perform usual daily activities) is presented as the mean percentage of activity impairment, calculated as 100*scale value of WPAI question 6 (between 0 and 10) / 10. WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity.
Time Frame: Baseline, Month 3, Month 6, Month 9
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: percentage of activity impairment
Arm/Group | Participants Receiving Anti-TNF for PsA
Number analyzed (Participants) | 120
percentage of activity impairment
  Baseline | 60.2 (19.2)
  Month 3: number analyzed (Participants) | 102
  Month 3 | 35.3 (23.7)
  Month 6: number analyzed (Participants) | 97
  Month 6 | 28.7 (20.9)
  Month 9: number analyzed (Participants) | 90
  Month 9 | 23.0 (20.6)
Statistical Analysis 1: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 9; Test type: Superiority; p < 0.001, Friedman test

5. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI) Score Up to Month 9
Description: The HAQ-DI is a participant-reported questionnaire. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide a total score ranging from 0 (no disability) to 3 (very severe, high-dependency disability).
Time Frame: Baseline, Month 3, Month 6, Month 9
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Anti-TNF for PsA
Number analyzed (Participants) | 120
units on a scale
  Baseline | 1.73 (0.50)
  Month 3: number analyzed (Participants) | 118
  Month 3 | 1.24 (0.65)
  Month 6: number analyzed (Participants) | 114
  Month 6 | 1.15 (0.63)
  Month 9: number analyzed (Participants) | 107
  Month 9 | 1.08 (0.59)
Statistical Analysis 1: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 3; Test type: Superiority; p < 0.001, Friedman test
Statistical Analysis 2: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 6; Test type: Superiority; p < 0.001, Friedman test
Statistical Analysis 3: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 9; Test type: Superiority; p < 0.001, Friedman test

6. Secondary Outcome: Percentage of Participants With American College of Rheumatology 20%, 50%, 70% (ACR20, ACR50, ACR70) Response at Month 9
Description: A participant is an ACR20, ACR50, or ACR70 responder if the following 3 criteria for improvement from Baseline are met:
  * ≥ 20%, ≥ 50%, or ≥ 70% improvement in tender joint count;
  * ≥ 20%, ≥ 50%, or ≥ 70% improvement in swollen joint count; and
  * ≥ 20%, ≥ 50%, or ≥ 70% improvement in at least 3 of the 5 following parameters:
    * Physician's global assessment of disease activity
    * Participant's global assessment of disease activity
    * Participant's assessment of pain
    * HAQ-DI
    * Acute phase reactant (erythrocyte sedimentation rate/C-reactive protein).
Time Frame: Month 9
Population: Participants with an assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Receiving Anti-TNF for PsA
Number analyzed (Participants) | 91
percentage of participants
  ACR20 Responder = No | 13.2
  ACR20 Responder = Yes | 86.8
  ACR50 Responder = No | 36.3
  ACR50 Responder = Yes | 63.7
  ACR70 Responder = No | 58.2
  ACR70 Responder = Yes | 41.8

7. Secondary Outcome: Disease Activity Score (DAS 28) Up to Month 9
Description: The DAS28 is a validated index of arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, C-reactive protein, and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10, with higher scores indicating higher disease activity. Participants were classified according to their scores as below:
  * DAS28 > 5.1 = High disease activity
  * DAS28 < 3.2 = Low disease activity
  * DAS28 < 2.6 = Remission
Time Frame: Baseline, Month 3, Month 6, Month 9
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Anti-TNF for PsA
Number analyzed (Participants) | 120
Participants
  Baseline: < 2.6 | 1
  Baseline: 2.6 to 3.2 | 6
  Baseline: 3.2 to 5.1 | 49
  Baseline: > 5.1 | 62
  Baseline: Missing | 2
  Month 3: < 2.6 | 32
  Month 3: 2.6 to 3.2 | 19
  Month 3: 3.2 to 5.1 | 34
  Month 3: > 5.1 | 16
  Month 3: Missing | 19
  Month 6: < 2.6 | 38
  Month 6: 2.6 to 3.2 | 29
  Month 6: 3.2 to 5.1 | 20
  Month 6: > 5.1 | 6
  Month 6: Missing | 27
  Month 9: < 2.6 | 49
  Month 9: 2.6 to 3.2 | 21
  Month 9: 3.2 to 5.1 | 15
  Month 9: > 5.1 | 4
  Month 9: Missing | 31

8. Secondary Outcome: Maastricht Ankylosing Spondylitis Enthesitis Scale (MASES) Up to Month 9
Description: For calculation of the enthesitis (tenderness) score, MASES was used in practice by the physicians. This scale takes into account the sites (first costochondral joint, seventh costochondral joint, posterior superior iliac spine, anterior superior iliac spine, iliac crest, fifth lumbar spinous process and proximal insertion of the Achilles tendon) and they scored from 0 to 13. Minimum tenderness score was 0; maximum tenderness score was 13.
Time Frame: Baseline, Month 3, Month 6, Month 9
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Anti-TNF for PsA
Number analyzed (Participants) | 119
units on a scale
  Baseline | 1.75 (2.37)
  Month 3: number analyzed (Participants) | 103
  Month 3 | 0.60 (1.50)
  Month 6: number analyzed (Participants) | 96
  Month 6 | 0.19 (0.76)
  Month 9: number analyzed (Participants) | 88
  Month 9 | 0.45 (1.50)
Statistical Analysis 1: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 3; Test type: Superiority; p < 0.001, Friedman test
Statistical Analysis 2: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 6; Test type: Superiority; p < 0.001, Friedman test
Statistical Analysis 3: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 9; Test type: Superiority; p < 0.001, Friedman test

9. Secondary Outcome: Dactylitis Score Up to Month 9
Description: A total of 20 digits were assessed as entire digits, looking for signs of tender dactylitis. Dactylitis is defined as a uniform swelling of the digits where the joints cannot be defined. Investigators entered scores between 0 (no swelling or pain) and 6 (most severe swelling and pain).
Time Frame: Baseline, Month 3, Month 6, Month 9
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Anti-TNF for PsA
Number analyzed (Participants) | 118
units on a scale
  Baseline | 0.47 (1.01)
  Month 3: number analyzed (Participants) | 103
  Month 3 | 0.15 (0.60)
  Month 6: number analyzed (Participants) | 95
  Month 6 | 0.06 (0.43)
  Month 9: number analyzed (Participants) | 88
  Month 9 | 0.03 (0.24)
Statistical Analysis 1: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 3; Test type: Superiority; p < 0.001, Friedman test
Statistical Analysis 2: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 6; Test type: Superiority; p < 0.001, Friedman test
Statistical Analysis 3: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 9; Test type: Superiority; p < 0.001, Friedman test

10. Secondary Outcome: Number of Swollen Joints Up to Month 9
Description: Twenty-eight joints were assessed and classified as swollen/not swollen by pressure and joint manipulation on physical examination. The presence of swelling is scored 1 and no swelling is 0; range of score is 0-28, with higher scores indicating more swollen joints.
Time Frame: Baseline, Month 3, Month 6, Month 9
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Participants Receiving Anti-TNF for PsA
Number analyzed (Participants) | 120
swollen joints
  Baseline | 4.91 (4.88)
  Month 3: number analyzed (Participants) | 97
  Month 3 | 1.99 (3.78)
  Month 6: number analyzed (Participants) | 90
  Month 6 | 0.39 (0.87)
  Month 9: number analyzed (Participants) | 84
  Month 9 | 0.54 (1.38)
Statistical Analysis 1: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 9; Test type: Superiority; p < 0.001, Friedman test

11. Secondary Outcome: Number of Tender Joints Up to Month 9
Description: Twenty-eight joints were assessed and classified as tender/not tender by pressure and joint manipulation on physical examination. The presence of tenderness is scored 1 and no tenderness is 0; range of score is 0-28, with higher scores indicating more tender joints.
Time Frame: Baseline, Month 3, Month 6, Month 9
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Participants Receiving Anti-TNF for PsA
Number analyzed (Participants) | 120
tender joints
  Baseline | 8.24 (8.22)
  Month 3: number analyzed (Participants) | 96
  Month 3 | 3.91 (6.98)
  Month 6: number analyzed (Participants) | 90
  Month 6 | 1.38 (2.41)
  Month 9: number analyzed (Participants) | 84
  Month 9 | 1.92 (4.14)
Statistical Analysis 1: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 3; Test type: Superiority; p < 0.001, Friedman test
Statistical Analysis 2: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 6; Test type: Superiority; p < 0.001, Friedman test
Statistical Analysis 3: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 9; Test type: Superiority; p < 0.001, Friedman test

12. Secondary Outcome: Levels of Rheumatoid Factor
Time Frame: Up to Month 9
Population: Since sufficient data could not be collected, this analysis was not performed.
Arm/Group | Participants Receiving Anti-TNF for PsA
Number analyzed (Participants) | 0

13. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR) Up to Month 9
Description: ESR values were measured as an inflammatory parameter. Low ESR values mean less inflammation.
Time Frame: Up to Month 9
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | Participants Receiving Anti-TNF for PsA
Number analyzed (Participants) | 96
mm/h
  Baseline: number analyzed (Participants) | 82
  Baseline | 6.46 (11.99)
  Month 3 | 14.71 (12.23)
  Month 6: number analyzed (Participants) | 87
  Month 6 | 14.28 (12.32)
  Month 9: number analyzed (Participants) | 84
  Month 9 | 15.65 (12.94)
Statistical Analysis 1: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 9; Test type: Superiority; p < 0.001, Friedman test

14. Secondary Outcome: C-reactive Protein (CRP) Up to Month 9
Description: CRP values were measured as an inflammatory parameter. Low CRP values mean less inflammation.
Time Frame: Baseline, Month 3, Month 6, Month 9
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Participants Receiving Anti-TNF for PsA
Number analyzed (Participants) | 118
mg/dL
  Baseline | 19.73 (48.06)
  Month 3: number analyzed (Participants) | 115
  Month 3 | 26.64 (18.63)
  Month 6: number analyzed (Participants) | 93
  Month 6 | 5.89 (10.20)
  Month 9: number analyzed (Participants) | 85
  Month 9 | 4.95 (7.85)

15. Secondary Outcome: Participant's Global Assessment of Disease Activity Visual Analog Scale (VAS) Up to Month 9
Description: A VAS was used to measure the participant's assessment of disease activity. For this assessment a 10-point scale was used (0: very well; 10: very poor).
Time Frame: Baseline, Month 3, Month 6, Month 9
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Anti-TNF for PsA
Number analyzed (Participants) | 120
units on a scale
  Baseline | 6.73 (1.63)
  Month 3: number analyzed (Participants) | 103
  Month 3 | 3.93 (2.76)
  Month 6: number analyzed (Participants) | 97
  Month 6 | 3.04 (1.82)
  Month 9: number analyzed (Participants) | 90
  Month 9 | 2.89 (2.15)
Statistical Analysis 1: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 3; Test type: Superiority; p < 0.001, Friedman test
Statistical Analysis 2: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 6; Test type: Superiority; p < 0.001, Friedman test
Statistical Analysis 3: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 9; Test type: Superiority; p < 0.001, Friedman test

16. Secondary Outcome: Physician's Global Assessment of Disease Activity VAS Up to Month 9
Description: A VAS was used to measure the physician's assessment of disease activity. For this assessment a 10-point scale was used (0: very well; 10: very poor).
Time Frame: Baseline, Month 3, Month 6, Month 9
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Anti-TNF for PsA
Number analyzed (Participants) | 120
units on a scale
  Baseline | 6.45 (1.35)
  Month 3: number analyzed (Participants) | 103
  Month 3 | 3.49 (2.16)
  Month 6: number analyzed (Participants) | 97
  Month 6 | 2.62 (1.54)
  Month 9: number analyzed (Participants) | 91
  Month 9 | 2.26 (1.74)
Statistical Analysis 1: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 3; Test type: Superiority; p < 0.001, Friedman test
Statistical Analysis 2: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 6; Test type: Superiority; p < 0.001, Friedman test
Statistical Analysis 3: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 9; Test type: Superiority; p < 0.001, Friedman test

17. Secondary Outcome: Participant's Assessment of Nocturnal Back Pain and Fatigue VAS Up to Month 9
Description: A VAS was used to measure the participant's assessment of nocturnal back pain and fatigue. For this assessment a 10-point scale was used (0: very well; 10: very poor).
Time Frame: Baseline, Month 3, Month 6, Month 9
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Anti-TNF for PsA
Number analyzed (Participants) | 120
units on a scale
  Baseline | 5.57 (2.50)
  Month 3: number analyzed (Participants) | 103
  Month 3 | 3.06 (2.84)
  Month 6: number analyzed (Participants) | 97
  Month 6 | 2.58 (2.24)
  Month 9: number analyzed (Participants) | 91
  Month 9 | 2.08 (2.08)
Statistical Analysis 1: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 3; Test type: Superiority; p < 0.001, Friedman test
Statistical Analysis 2: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 6; Test type: Superiority; p < 0.001, Friedman test
Statistical Analysis 3: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 9; Test type: Superiority; p < 0.001, Friedman test

18. Secondary Outcome: Participant's Assessment of Total Back Pain VAS Up to Month 9
Description: A VAS was used to measure the participant's assessment of back pain. For this assessment a 10-point scale was used (0: very well; 10: very poor).
Time Frame: Baseline, Month 3, Month 6, Month 9
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Anti-TNF for PsA
Number analyzed (Participants) | 120
units on a scale
  Baseline | 5.25 (2.64)
  Month 3: number analyzed (Participants) | 103
  Month 3 | 3.28 (2.46)
  Month 6: number analyzed (Participants) | 97
  Month 6 | 2.47 (2.22)
  Month 9: number analyzed (Participants) | 91
  Month 9 | 2.22 (2.16)
Statistical Analysis 1: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 3; Test type: Superiority; p < 0.001, Friedman test
Statistical Analysis 2: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 6; Test type: Superiority; p < 0.001, Friedman test
Statistical Analysis 3: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 9; Test type: Superiority; p < 0.001, Friedman test

19. Secondary Outcome: Participant's Assessment of Pain and Fatigue VAS Up to Month 9
Description: A VAS was used to measure the participant's assessment of pain and fatigue. For this assessment a 10-point scale was used (0: very well; 10: very poor).
Time Frame: Baseline, Month 3, Month 6, Month 9
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Anti-TNF for PsA
Number analyzed (Participants) | 120
units on a scale
  Baseline | 6.37 (1.75)
  Month 3: number analyzed (Participants) | 103
  Month 3 | 4.31 (6.93)
  Month 6: number analyzed (Participants) | 97
  Month 6 | 2.91 (2.17)
  Month 9: number analyzed (Participants) | 91
  Month 9 | 2.67 (2.45)
Statistical Analysis 1: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 3; Test type: Superiority; p < 0.001, Friedman test
Statistical Analysis 2: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 6; Test type: Superiority; p < 0.001, Friedman test
Statistical Analysis 3: Comparison: Participants Receiving Anti-TNF for PsA; Baseline vs. Month 9; Test type: Superiority; p < 0.001, Friedman test

20. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Discontinuations Due to Treatment-Related Adverse Events (AEs) Up to Month 9
Description: Number of participants with any serious adverse event (SAE) occurring during treatment with anti-TNF agents and/or participants who discontinued treatment due to SAEs or AEs which were caused by the treatment with anti-TNF agents during the course of treatment. An SAE is defined as an event that: results in the death; is life-threatening; results in an admission to the hospital or prolongation of hospitalization; is a congenital anomaly; results in a condition that substantially interferes with the activities of daily living of a study subject; is an important medical event according to the Investigator.
Time Frame: Up to Month 9
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Anti-TNF for PsA
Number analyzed (Participants) | 120
Participants
  Any SAE | 1
  Discontinuations | 0

ADVERSE EVENTS:
Time Frame: Up to Month 9
Description: SAEs were collected and reported; per protocol, non-serious AE data was not collected for this observational study.
Arm/Group | Participants Receiving Anti-TNF for PsA
Serious Adverse Events (participants affected / at risk) | 1/120
Other Adverse Events (participants affected / at risk) | 0/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Receiving Anti-TNF for PsA (N=120)
Tuberculosis of genitourinary system (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.